CLINICAL TRIAL: NCT04685252
Title: Investigating a Probiotic on Mothers' Mood and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 19.16.NRC
Record Dates: First submitted 2020-12-16; First posted 2020-12-28 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Perinatal Problems; Mood Change; Stress-related Problem
Keywords: probiotic; mood; stress; perinatal
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Individually unique coding for each stickpack
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Partum and Post-Partum (BL) NCC3001 (Experimental): One stickpack containing probiotic strain (BL) NCC3001, dissolved and consumed oral daily over a period of 6 months; 3 months pre- and post-partum.
  Interventions: Other: (BL) NCC3001
- Placebo Control (Placebo Comparator): One Placebo stickpack containing maltodextrin, dissolved and consumed oral daily over a period of 6 months; 3 months pre- and post-partum.
  Interventions: Other: Placebo
- Post-Partum (BL) NCC3001 (Crossover Arm) (Experimental): One Placebo stickpack containing maltodextrin, dissolved and consumed oral daily for 3 months during pre-partum, followed with switch to one stickpack containing probiotic strain (BL) NCC3001, dissolved and consumed oral daily for 3 months post-partum.
  Interventions: Other: (BL) NCC3001; Other: Placebo

INTERVENTIONS:
Other: (BL) NCC3001 — Probiotic strain (BL) NCC3001 packed in stickpack, to be consumed daily.
  Other Names: Bifidobacterium longum (BL) NCC3001
  Arms: Post-Partum (BL) NCC3001 (Crossover Arm); Pre-Partum and Post-Partum (BL) NCC3001
Other: Placebo — Matching placebo containing maltodextrin packed in stickpack, to be consumed daily.
  Other Names: Maltodextrin
  Arms: Placebo Control; Post-Partum (BL) NCC3001 (Crossover Arm)

SUMMARY:
This is a randomized, placebo-controlled, double-blind, 3 parallel-arm study in pregnant women aged 21 years old and above. The study aims to assess changes in perinatal mood and stress when administering a probiotic starting from either the 3rd trimester (i.e 28-32 weeks of gestational age) or immediately after birth, until 12 weeks post-partum.

DETAILED DESCRIPTION:
To date, limited evidence is available for nutritional interventions in the role of modulation of perinatal mood and stress, even less so for probiotics. The probiotic strain Bifidobacterium longum (BL) NCC3001 has previously been shown to normalize anxiety-like behavior in preclinical models and to reduce feelings of low mood and emotional reaction to fearful stimulus in human adults with irritable bowel syndrome (IBS). The strain is also considered safe and has previously been administered to pregnant and lactating women as well as infants. Therefore, the study aims to evaluate the effect of probiotic (BL) NCC3001 on mood and stress levels during the perinatal period.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 21 years-old or above at recruitment
* Willing and able to provide written informed consent
* Gestational age of 28-32 weeks at Randomization
* Singleton pregnancy at Recruitment
* Able to respond to questionnaires in English
* Hospital Anxiety and Depressive Scale (HADS) score of ≥ 5 (out of 21) for either subscale to indicate some general feelings of low mood and/or stress at screening
* Intention to breastfeed

Exclusion Criteria:

* Not willing and/or not able to comply with the study procedures and requirements
* Food allergy
* Has taken probiotic supplements in the period of 4 weeks prior to screening
* Has received pharmacological treatment for anxiety and/or depression in the period of 12 weeks prior to recruitment
* Major complications during pregnancy e.g., pre-eclampsia, gestational diabetes requiring insulin intervention, severe intra-uterine growth restriction (IUGR), fetal anomalies that in the opinion of the investigator may interfere with the pregnancy and participation in the clinical trial
* Pre-existing medical conditions e.g., hypertension, diabetes mellitus, thyroid diseases, autoimmune diseases such as Systemic Lupus Erythematosus, antiphospholipid syndrome and other major chronic illness that in the opinion of the investigator may interfere with the pregnancy and participation in the clinical trial
* Active participation in another clinical trial or on-going observational study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 184 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Change in EPDS score | through study completion, an average of 6 months
  Measure change in trend of Edinburgh Postnatal Depression Scale (EPDS)
Change in STAI score | through study completion, an average of 6 months
  Measure change in trend of State Trait Anxiety Inventory (STAI)

SECONDARY OUTCOMES:
Risk of EPDS score ≥ 13 | through study completion, an average of 6 months
  Number of subjects reaching Edinburgh Postnatal Depression Scale (EPDS) ≥ 13
Salivary Cortisol | through study completion, an average of 6 months
  Measure change in the salivary cortisol levels
Parenting stress | 12 weeks post-partum
  Measured by the Parenting Stress Index (PSI) questionnaire
Sleep quality | 36 weeks pre-partum and 12 weeks post-partum
  Measured by the Pittsburgh sleep quality index (PSQI)
Microbiota composition of stool | Baseline to 12 weeks post-partum
  Measure changes in the microbiota composition and probiotic strain colonization
Gastrointestinal comfort | through study completion, an average of 6 months
  Measure changes in Gastrointestinal symptom rating score (GSRS)
Breastfeeding practices | Baseline and post-partum (9 days, 4 weeks, 8 weeks and 12 weeks)
  Measure changes in Early Feeding Questionnaire (EFQ)
Anxiety and depressive symptoms | Baseline and at 12 weeks post-partum
  Measured by change in Hospital anxiety and depression scale (HADs)
Digital assessments of stress | Throughout the entire study
  Change in stress index measured using ANURA application

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fries, PhD., Study Chair — NESTLE RESEARCH
Locations (1):
- Singapore Institute for Clinical Sciences, A*STAR Research Entities, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toh MPS, Yang CY, Lim PC, Loh HLJ, Bergonzelli G, Lavalle L, Mardhy E, Samuel TM, Suniega-Tolentino E, Silva Zolezzi I, Fries LR, Chan SY. A Probiotic Intervention With Bifidobacterium longum NCC3001 on Perinatal Mood Outcomes (PROMOTE Study): Protocol for a Decentralized Randomized Controlled Trial. JMIR Res Protoc. 2023 Apr 5;12:e41751. doi: 10.2196/41751. PMID 37018024